CLINICAL TRIAL: NCT04013438
Title: Duration of Estrogen for Luteal Phase in Pregnant Women Undergone Frozen Embryo Transfer Cycles- Randomized Controlled Trials Phase III
Brief Title: Luteal Phase Support During Frozen Embryo Transfer Cycle
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Royan, Female Infertility,LPS
Record Dates: First submitted 2019-05-28; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-05

CONDITIONS: Infertility, Female; Frozen Embryo Transfer
Keywords: Ongoing pregnancy rate; Estrogen; Frozen embryo transfer; Luteal phase support
MeSH Terms: conditions — Infertility, Female | interventions — IDS 89 Sabal serrulata extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FET cycle, discontinue estradiol after 6 gestational weeks (Experimental): In patients 35 days after embryo transfer and observation of gestational sac with heart beat (6 weeks of pregnancy) by ultrasound, exogenous estrogen will discontinued while progesterone will remain daily use until twelfth week of pregnancy.
  Interventions: Drug: Strogen
- FET cycle, continue estradiol till 12 gestational weeks (Active Comparator): Control group receive 6 mg oral estrogen and 100 mg intramuscularly progesterone until 12 week of pregnancy.
  Interventions: Drug: Strogen

INTERVENTIONS:
Drug: Strogen — The OCP-LD begins in 2 to 3 days of the last menstrual cycle and then 500 μgr/d GnRH-a will received on day 17 for fourteen days. Then in 2-3 days of the next menstrual cycle, GnRH-a reduced to 200 μgr/d dose. the patients will receive 6 mg oral that will be continued for 14 days and during this time endometrium thickness evaluated by vaginal ultrasonography. If endometrial thickness is estimated ≥7mm, intramuscularly progesterone 100 mg/d will be started. After the onset of progesterone (days 17 to 18 cycles) frozen embryos transferred. Control group receive 6 mg oral estrogen and 100 mg intramuscularly progesterone until 12 week of pregnancy. The levels of maternal estrogen and progesterone was measured at the time of the starting day of progesterone (day 15), the day of embryo transfer, 6 and 12 weeks of pregnancy.
  Other Names: estradiol till 12 gestational weeks
  Arms: FET cycle, continue estradiol till 12 gestational weeks
Drug: Strogen — The OCP-LD begins in 2 to 3 days of the last menstrual cycle and then 500 μgr/d GnRH-a will received on day 17 for fourteen days. Then in 2-3 days of the next menstrual cycle, GnRH-a reduced to 200 μgr/d dose. the patients will receive 6 mg oral that will be continued for 14 days and during this time endometrium thickness evaluated by vaginal ultrasonography. If endometrial thickness is estimated ≥7mm, intramuscularly progesterone 100 mg/d will be started. After the onset of progesterone (days 17 to 18 cycles) frozen embryos transferred. In patients 35 days after embryo transfer and observation of gestational sac with heart beat (6 weeks of pregnancy) by ultrasound, exogenous estrogen will discontinued while progesterone will remain daily use until twelfth week of pregnancy. The levels of maternal estrogen and progesterone was measured at the time of the starting day of progesterone (day 15), the day of embryo transfer, 6 and 12 weeks of pregnancy.
  Other Names: estradiol till 6 gestational weeks
  Arms: FET cycle, discontinue estradiol after 6 gestational weeks

SUMMARY:
We aimed to decrease quantity of exogenous estrogen and evaluated the success rate of ongoing pregnancy in women undergone artificial FET who have a surplus embryos at previous fertility treatment cycles.

In this study, endometrial prepared with standard long GnRH protocol and for luteal phase support patients received 6 mg oral E2 and intramuscularly P 100 mg/d and embryos on day 2-3 were transferred. Control group continued E2 until 12 week of pregnancy, while for cases after identify gestational sac with heart beat (the 6 week of pregnancy) by vaginal ultrasonography, E2 will discontinued.

DETAILED DESCRIPTION:
Approval Status: Confirmed Approval reference Number: IR.ACECR.ROYAN.REC.1395.70 Board Name: Ethics committee of Royan infertility institute Board Affiliation: Reza Samani Phone: +982122305236 Email: samani@royaninstitute.org

Yes Health, Treatment and Medical Education Ministry: Iran

Hormones replace therapy (Artificial) is a method for endometrium preparation and embryo transfer. In this protocol for decrease of spontaneous ovulation, exogenous estrogen began in 2-3 days on follicular phase of the menstrual cycle which continue about 10 to 14 days. In the following luteal phase support by progesterone begins on 14 to 16 days of cycles. The luteal phase is supported with different dose and duration of estradiol (E2) and progesterone (P) until 8-12 week of pregnancy. Studied reported a higher risk of thromboembolism in pregnant women that using exogenous estrogen. Also, excess estrogen might be resulted fetus congenital anomalies, low birth weight and increased susceptibility to breast cancer in female fetuses. On the other hands, it seems placenta in early pregnancy duration synthesize estrogen and this time estrogen sufficient as a product of progesterone metabolism. We aimed to decrease quantity of exogenous estrogen and evaluated the success rate of ongoing pregnancy in women undergone artificial FET who have a surplus embryos at previous fertility treatment cycles.

In this study, endometrial prepared with standard long GnRH protocol and for luteal phase support patients received 6 mg oral E2 and intramuscularly P 100 mg/d and embryos on day 2-3 were transferred. Control group continued E2 until 12 week of pregnancy, while for cases after identify gestational sac with heart beat (the 6 week of pregnancy) by vaginal ultrasonography, E2 will discontinued.

The level of maternal estrogen and progesterone measured at progesterone days (day 15), the day of embryo transfer, 6 and 12 weeks of pregnancy.

This study is a randomized clinical trial to investigate the duration of estrogen for luteal phase in pregnant women undergone frozen embryo transfer cycles- Randomized controlled trials phase III. The study protocol is approved by the Ethics Committee (Institutional Review Board) of Royan institute and all participants provide informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with surplus embryos undergone infertility treatment cycles (e.g. OHSS, inadequate endometrium, surplus frozen embryo from any cause)
2. Age 21-37 years
3. Normal BMI (18.5 <BMI <30)
4. IVF / ICSI or IVF or ICSI cycles with antagonists or agonists protocols
5. Frozen embryos on 2-3 days

Exclusion Criteria:

1. Endometrial thickness ≤7mm
2. Egg Donors
3. Surrogacy
4. Male factor infertility with azoospermia
5. Age <37 years old
6. Hydrosalpinx
7. Uterine anomalies
8. Myoma with a compression effect or submocusa myoma
9. PGD
10. Blastocyst embryo transfer, ZIFT and GIFT

Ages: 21 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate after frozen embryo transfer | ≥20 weeks of gestational age
  Ongoing pregnancy was defined when the pregnancy had completed ≥20 weeks of gestation.

SECONDARY OUTCOMES:
Maternal serum estrogen level | The start day of using progesterone for luteal support in FET cycle (day 15 after onset estradiol), the day of embryo transfer (approximately 17-18 days after onset estradiol), 6 and 12 weeks of gestational age
  Maternal serum estrogen level
Maternal serum progesterone level | The start day of using progesterone for luteal support in FET cycle (day 15 after onset estradiol), the day of embryo transfer (approximately 17-18 days after onset estradiol), 6 and 12 weeks of gestational age
  Maternal serum progesterone level

CONTACTS AND LOCATIONS:
Locations (1):
- Royan Institute, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ghaffari F, Chekini Z, Vesali S. Duration of estradiol supplementation in luteal phase support for frozen embryo transfer in hormone replacement treatment cycles: a randomized, controlled phase III trial. Arch Gynecol Obstet. 2022 Mar;305(3):767-775. doi: 10.1007/s00404-021-06173-w. Epub 2021 Sep 24. PMID 34561715